CLINICAL TRIAL: NCT04928365
Title: Open Prospective Clinical Trial to Develop the Computer Software (Intelligent Prognostic System) for Predicting the Efficacy of Anti-PD-1 Immunotherapy of Melanoma Patients in Routine Practice
Brief Title: Evaluation of Cytokine Biomarkers in Melanoma Patients During Immunotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Responsible Party: Principal Investigator, Irina Mikhaylova, Principal investigator, Blokhin's Russian Cancer Research Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Cytokim-01
Record Dates: First submitted 2021-06-07; First posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced melanoma patients (Other)
  Interventions: Drug: Anti-PD-1 monoclonal antibody
- Stage III and IV melanoma patients after radical surgery (Other)
  Interventions: Drug: Anti-PD-1 monoclonal antibody

INTERVENTIONS:
Drug: Anti-PD-1 monoclonal antibody — Anti-PD-1 therapy

SUMMARY:
Open prospective clinical trial to develop the computer software (Intelligent prognostic system) for predicting the efficacy of anti-PD-1 immunotherapy of melanoma patients in routine practice

ELIGIBILITY:
Inclusion Criteria:

1. Morphological verification of cutaneous melanoma. Verification of metastases is not necessary
2. ECOG 0-1
3. Age of patients - 18 years and older
4. No prior chemotherapy, immunotherapy, radiation or hormonal therapy
5. Adequate contraception for women of childbearing age
6. Written consent of the patient to participate in the study

Exclusion Criteria:

1. Non-compliance with the previously listed criteria
2. Pregnancy and breastfeeding
3. Therapy with systemic corticosteroids and/or other immunosuppressants within 4 weeks before the screening or a high probability of the need for their use during the study for the treatment of intercurrent pathology
4. History of another malignancy other than the study indication under this trial within 5 years of study enrollment. Does not apply to subjects who underwent successful definitive resection of basal or squamous cell carcinoma of the skin, in situ cervical cancer, in situ breast cancer, or other in situ cancers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2023-03-25 (Estimated)

PRIMARY OUTCOMES:
Overall survival | up to 12 months
Progression free survival | up to 12 months

SECONDARY OUTCOMES:
Cytokine profile | up to 12 months
  IL-2, IL-6, IL-7, IL-8, IL-10, IL-12p70, IL-22, (IFN)-α2, IFN-γ, NFβ/Lymphotoxin-α(LTA), MCP-1/CCL2,IP-10/CXCL10, MIG/CXCL9, GM-CSF, PDGF-AA, PDGF-AB/BB, VEGF-A

CONTACTS AND LOCATIONS:
Locations (1):
- N.N. Blokhin Russian Cancer Research Center, Kashirskoye shosse 23, Moscow, Russia